CLINICAL TRIAL: NCT03013010
Title: A Randomized, Controlled, Multicenter Study to Compare Preoperative Radiochemotherapy With Preoperative Chemotherapy in Patients With Locally Advanced Gastric or Esophagogastric Junction Adenocarcinoma (PREACT Study)
Brief Title: PREACT Study: Locally Advanced Gastric Cancer, Chemoradiotherapy vs. Chemotherapy Followed by D2 Surgery and Adjuvant Chemotherapy
Acronym: PREACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Cancer Hospital, China (Other)
Collaborators: Fudan University (Other); Ruijin Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Huadong Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUSCC-LAGCCS002
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Stomach Neoplasm; GastroEsophageal Cancer; Adenocarcinoma; Locally Advanced Cancer; Chemoradiation
Keywords: Randomized; Open Label; Multicenter
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma | interventions — S 1 (combination); Chemoradiotherapy; Gastrectomy; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preoperative radiochemotherapy (Experimental): 1 cycle preoperative chemotherapy with S-1(Tegafur-Gimeracil-Oteracil Potassium)+ oxaliplatin.
  5 weeks preoperative chemoradiotherapy.
  1 cycle preoperative chemotherapy with S-1(Tegafur-Gimeracil-Oteracil Potassium)+ oxaliplatin.
  Gastric resection. 3 cycles adjuvant chemotherapy with S-1(Tegafur-Gimeracil-Oteracil Potassium)+ oxaliplatin.
  Interventions: Drug: Tegafur-Gimeracil-Oteracil Potassium; Radiation: Chemoradiotherapy; Procedure: Gastric resection; Drug: Oxaliplatin
- Preoperative chemotherapy (Active Comparator): 3 cycles preoperative chemotherapy with S-1(Tegafur-Gimeracil-Oteracil Potassium)+ oxaliplatin.
  Gastric resection. 3 cycles adjuvant chemotherapy with S-1(Tegafur-Gimeracil-Oteracil Potassium)+ oxaliplatin.
  Interventions: Drug: Tegafur-Gimeracil-Oteracil Potassium; Procedure: Gastric resection; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Tegafur-Gimeracil-Oteracil Potassium — The dose of S-1 is according to body-surface area (BSA): patients with a BSA of less than 1.25 m2 received 80 mg daily; those with a BSA of 1.25 m2 or more but less than 1.5 m2 received 100 mg daily; and those with a BSA of 1.5 m2 or more received 120 mg daily. oxaliplatin 130mg/m2, intravenously, on day 1.
  Other Names: S-1
Radiation: Chemoradiotherapy — Chemotherapy: S-1 40-60mg/m2 orally, oral tablet twice daily, days 1-5 of each week of radiotherapy.
  Radiotherapy: 45 Gy of radiation in 25 fractions, five days per week for five weeks.
  Other Names: radiochemotherapy
  Arms: Preoperative radiochemotherapy
Procedure: Gastric resection — A standard D2 gastrectomy was recommended. The type of gastrectomy performed depended on the location and extent of the primary lesion. For middle third tumors, the gastric margin was recommended to be more than 5 cm, and a total gastrectomy was performed. For lower third tumors, a 2 cm duodenal margin was recommended and a subtotal or total gastrectomy was considered. For upper third tumors, a 3 cm esophageal margin was recommended and a total gastrectomy or esophagogastrectomy was performed. Billroth I or Roux-en-y gastrojejunostomy was performed for distal gastrectomy patients, Roux-en-y esophagojejunostomy was performed for total gastrectomy patients.
  Other Names: Gastrectomy
Drug: Oxaliplatin — The dose of oxaliplatin is according to body-surface area (BSA): 130mg/m2, intravenously, on day 1.

SUMMARY:
Although the incidence of gastric cancer has been substantially declining for several decades, it is still the sixth most common cancer and the fourth most frequent cause of cancer death worldwide. Surgery is still the only curative option for gastric cancer. However, most patients are unable to undergo surgery because of late stage, unresectable disease. The prognosis for these patients is very poor. Although the Magic trial showed that perioperative chemotherapy can increase the rate of curative surgery and significantly improve overall survival in patients with operable gastric or lower esophageal adenocarcinomas, no pCR events were reported in this trial. The intervention arm in PREACT consists of pre-operative chemotherapy, pre-operative radiochemotherapy, surgery and post-operative chemotherapy. The control arm consists of pre-operative chemotherapy, surgery, and post-operative chemotherapy. The primary purpose of PREACT is to investigate whether the addition of radiochemotherapy to chemotherapy is superior to chemotherapy alone in the pre-operative setting in improving disease free survival in patients with locally advanced gastric or esophagogastric junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* Female and male
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Life expectancy >=6 months
* Histologically proven adenocarcinoma of the stomach or gastroesophageal junction (GEJ) (excluding Siewert I) that is: Stage IIB (T3N1 only), IIIA (T2N3 not eligible), IIIB, and IIIC, i.e. T3 - T4a and node positive, or T4b and/ or node positive, according to American Joint Committee on Cancer (AJCC) 7th edition
* Considered operable following initial staging investigations or after pre-operative therapy Disease which can be radically treated with radiotherapy to 45 Gy with standard fractionation
* Adequate organ function defined as follows:
* Bone marrow: Haemoglobin >=90 g/L, Absolute neutrophil count (ANC) >=1.5 x 109 /L, Platelet count >=100 x 109 /L; Hepatic: Serum bilirubin <=1.5 x upper limit of normal, aspartate aminotransferase (AST) and/or alanine transaminase (ALT) <=2.5 x upper limit of normal; Renal: Serum creatinine <=1.0 x upper limit of normal
* Patients are willing to obey the treatment and provide blood and tissue specimens
* Written informed consent obtained before randomization

Exclusion Criteria:

* Pregnant or lactating females or female patients of childbearing potential who have not been surgically sterilized or are without adequate contraceptive measures
* Sexually active males or females refuse to practice contraception during the study until 30 days after end of study
* Evidence of metastatic disease
* Prior chemotherapy or radiotherapy
* Patients with a past history of cancer in the 5 years before randomization except for the squamous or basal cell carcinoma of the skin that has been effectively treated, and carcinoma in situ of the cervix that has been treated by operation
* Patients with other significant underlying medical conditions that may be aggravated by the study treatment or are not controlled
* Patients with central nervous system(CNS) disorder or peripheral nervous system disorder or psychiatric disease
* Known history of uncontrolled or symptomatic angina, uncontrolled arrhythmias and hypertension, or congestive heart failure, or cardiac infarction within 6 months prior to study enrollment, or cardiac insufficiency
* Concurrent severe infection
* Severe gastrointestinal bleeding, gastrointestinal perforation
* Unable to swallow
* Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical disorder that would interfere with the subject's safety
* Known hypersensitivity reaction or metabolic disorder to S-1or oxaliplatin
* Renal impairment (GFR <=50ml/min)
* Linitis plastica

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Disease free survival | up to 3 years

SECONDARY OUTCOMES:
Overall survival | up to 3 years
Surgical complete resection rate (R0) | at the time of surgery
Pathological response rate | at the time of surgery
Proportion of patients with toxicities | up to 3 years
Proportion of patients with surgery-related complication | at the time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ya-nong Wang, M.D., Principal Investigator — Fudan University; Zhen Zhang, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Liu X, Jin J, Cai H, Huang H, Zhao G, Zhou Y, Wu J, Du C, Long Z, Fang Y, Ma M, Li G, Zhou M, Yin J, Zhu X, Zhu J, Sheng W, Huang D, Zhu H, Zhang Z, Lu Q, Xie L, Zhang Z, Wang Y. Study protocol of a randomized phase III trial of comparing preoperative chemoradiation with preoperative chemotherapy in patients with locally advanced gastric cancer or esophagogastric junction adenocarcinoma: PREACT. BMC Cancer. 2019 Jun 20;19(1):606. doi: 10.1186/s12885-019-5728-8. PMID 31221115
- [Derived] Liu X, Cai H, Sheng W, Huang H, Long Z, Wang Y. microRNAs expression profile related with response to preoperative radiochemotherapy in patients with locally advanced gastric cancer. BMC Cancer. 2018 Oct 29;18(1):1048. doi: 10.1186/s12885-018-4967-4. PMID 30373600